CLINICAL TRIAL: NCT05631015
Title: Development and Validation of Gastroscopy Surveillance Recommendations Based on Natural Language Processing for Patients With Gastric Cancer and Precancerous Diseases
Brief Title: Artificial Intelligence for Determination of Gastroscopy Surveillance Intervals
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xiuli Zuo (Other)
Responsible Party: Sponsor-Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Organization: Shandong University (Other)
Other Study IDs: 2022-SDU-QILU-G008
Record Dates: First submitted 2022-11-19; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Helicobacter Pylori Infection; Atrophic Gastritis; Intestinal Metaplasia; Low Grade Intraepithelial Neoplasia; High Grade Intraepithelial Neoplasia; Early Gastric Cancer; Gastric Cancer
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Artificial Intelligence support decision group: According the endoscopic reports and pathological reports, the decision support system recognise patients' disease types and grades, and generate guidelines based survilliance or treatment recommendations.
  Interventions: Other: AI recongnize disease and generate recommendations

INTERVENTIONS:
Other: AI recongnize disease and generate recommendations — According the endoscopic reports and pathological reports, the decision support system recognise patients' disease types and grades, and generate guidelines based survilliance or treatment recommendations.

SUMMARY:
The purpose of this study is to develop and validate a clinical decision support system based on automated algorithms. This system can use natural language processing to extract data from patients' endoscopic reports and pathological reports, identify patients' disease types and grades, and generate guidelines based follow-up or treatment recommendations

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 80 years
* Patients underwent endoscopic examination

Exclusion Criteria:

* Patients with the contraindications to endoscopic examination
* Patients with imcomplete examination information
* Patients undergo endoscopy for therapy
* Patients have history of upper gastrointestinal surgery
* Patients with duodenal or Laryngeal neoplasms
* Patients with gastrointestinal submucosal tumor

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who came to Qilu Hospital of Shandong University and received endoscopy examination but not therapeutic endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of gastric diseases with deep learning algorithm | 12 month
  The diagnostic accuracy of gastric diseases with deep learning algorithm
The accuracy of recommentions for different disease with deep learning algorithm | 12 month
  The accuracy of recommentions for different disease with deep learning algorithm

SECONDARY OUTCOMES:
The diagnostic sensitivity of gastric diseases with deep learning algorithm | 12 month
  The diagnostic sensitivity of gastric diseases with deep learning algorithm
The diagnostic specificity of gastric diseases with deep learning algorithm | 12 month
  The diagnostic specificity of gastric diseases with deep learning algorithm
The diagnostic positive predictive value of gastric diseases with deep learning algorithm | 12 month
  The diagnostic positive predictive valu of gastric diseases with deep learning algorithm
The diagnostic negative predictive value of gastric diseases with deep learning algorithm | 12 month
  The diagnostic negative predictive value of gastric diseases with deep learning algorithm
The F-score of gastric diseases with deep learning algorithm | 12 month
  The F-score of gastric diseases with deep learning algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China